CLINICAL TRIAL: NCT04426708
Title: An Open-Label, Paralleled Study of the Pharmacokinetics of HMS5552 Following a Single Oral Dose in Mild and Moderate Hepatic Impaired Subjects and Matched Healthy Volunteers
Brief Title: A Clinical Study to Access the Pharmacokinetics of HMS5552 in Hepatic Impaired Subjects and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMM0109
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dorzagliatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild hepatic impaired subjects (A) (Experimental): Mild hepatic impaired subjects: to receive a single dose of HMS5552 ( 25mg ) tablet orally
  Interventions: Drug: HMS5552
- Moderate hepatic impaired subjects (B) (Experimental): Moderate hepatic impaired subjects: to receive a single dose of HMS5552 ( 25mg ) tablet orally
  Interventions: Drug: HMS5552
- Healthy volunteers (C) (Experimental): Matched healthy volunteers: to receive a single dose of HMS5552 ( 25mg ) tablet orally
  Interventions: Drug: HMS5552

INTERVENTIONS:
Drug: HMS5552 — single dose of HMS5552 25mg

SUMMARY:
The objectives of this study is to access the pharmacokinetics and safety of HMS5552 in single dose in mild and moderate hepatic impaired subjects and matched healthy adult subjects.

DETAILED DESCRIPTION:
This is an open-label and paralleled study with single oral dose of HMS5552 given to hepatic impaired subjects and matched healthy volunteers.

The primary objective is to access the pharmacokinetic profiles of HMS5552 in 25 mg dose in hepatic impaired subjects and (gender, age and BMI) matched healthy adult subjects.

The secondary objective is to characterize the safety profiles of HMS5552 in single dose in hepatic impaired subjects.

The subjects include mild hepatic impaired subjects (A group), moderate hepatic impaired subjects (B group), and healthy subjects (C Group) matched with hepatic impaired subjects in gender, age and BMI. The number of subjects in each group was no less than 8, and no less than 3 subjects in each gender.

ELIGIBILITY:
Inclusion Criteria:

* For hepatic impaired subjects:

  1. Male and female subjects between ages of 18 and 65 years, no less than 3 subjects in each gender.
  2. Body weight≥50kg for male and ≥45kg for female； BMI: 18.5~30 kg/m2
  3. ALT>2×normal upper limit (ULN), or TBiL>1.5×ULN, or diagnosed cirrhosis. The related clinical manifestations have been stable for 4-12 weeks, and Child-Pugh score is in grade A or B:

     A= mild liver damage (Group A): Child-Pugh 5-6; B= moderate liver damage (Group B): Child-Pugh 7-9;
  4. Willing to sign the informed consent form (ICF) and take reliable contraceptive measures within 6 months after taking the last dose of study drug;
  5. Willing to adhere to the protocol requirement.
* For healthy volunteers:

  1. Male and female subjects between ages of 18 and 65 years, no less than 3 subjects in each gender;
  2. Body weight≥50kg for male and ≥45kg for female； BMI: 18.5~30 kg/m2;
  3. Gender, age (±5 years) and BMI (±15%) matched with corresponding subject in hepatic impaired group;
  4. Normal physical conditions, vital signs,12 lead ECG and laboratory recording;
  5. Willing to sign the informed consent form (ICF) and take reliable contraceptive measures within 6 months after taking the last dose of study drug;
  6. Willing to adhere to the protocol requirement.

Exclusion Criteria:

* Subjects with impaired hepatic function cannot be enrolled if they meet one of the following criteria:

  1. Liver cancer, liver transplantation, liver failure, autoimmune liver disease, biliary cirrhosis, or drug-induced liver damage;
  2. History of allergy;
  3. Investigators adjudicate subjects have surgery that may affect drug absorption, distribution, metabolism or excretion;
  4. In addition to diseases and complications of impaired hepatic function, investigator adjudicate subjects have clinically meaningful or unstable diseases or complications of central nervous system, cardiovascular system, digestive system, endocrine system, respiratory system, urinary system, blood system, mental disease, or malignant tumor, etc;
  5. Abnormal of ECG performance or laboratory recording during screening;
  6. Family history of QT prolongation syndrome;
  7. History of hepatic encephalopathy or hepatic coma within 6 months before screening;
  8. More than 5 cigarettes per day within 3 months before screening;
  9. Alcohol addicts;
  10. History of drug abuse
* Healthy subjects cannot be enrolled if they meet one of the following criteria:

  1. History of allergy;
  2. Investigators adjudicate subjects have surgery that may affect drug absorption, distribution, metabolism or excretion;
  3. Investigator adjudicate subjects have clinically meaningful or unstable diseases or complications of central nervous system, cardiovascular system, digestive system, endocrine system, respiratory system, urinary system, blood system, mental disease, or malignant tumor, etc;
  4. Abnormal of ECG performance or laboratory recording during screening;
  5. Family history of QT prolongation syndrome;
  6. Severe infection, severe trauma or major surgery judged by investigator within 3 months before screening;
  7. More than 5 cigarettes per day within 3 months before screening;
  8. Alcohol addicts;
  9. History of drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of Cmax; | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of AUClast; | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of AUCinf; | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.

SECONDARY OUTCOMES:
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of Cmax,u | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of AUClast,u | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of AUCinf,u | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of Tmax ; | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of T1/2; | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of CL/F; | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of Vz/F; | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of fu; | Up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hour post-dose.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No